CLINICAL TRIAL: NCT05721781
Title: Reducing Risk for Infective Endocarditis (IE): A Randomized Trial of a Professional Scaling and Oral Hygiene Instruction Intervention to Reduce Tooth Brushing-Associated Bacteremia
Brief Title: Reducing Risk for Infective Endocarditis
Acronym: PIE-B
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00092954
Record Dates: First submitted 2023-01-31; First posted 2023-02-10 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Bacteremia; Infective Endocarditis
Keywords: Oral Hygiene; Oral Bacteria; Gingival inflammation
MeSH Terms: conditions — Bacteremia; Endocarditis; Gingivitis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants receiving a dental cleaning and oral hygiene instruction (Experimental): Participants randomized to this arm will receive a standard dental cleaning and education on proper toothbrushing and flossing technique and asked to follow these toothbrushing and flossing techniques for the duration of the study period. They will receive periodic phone call reminders to maintain these practices during the study period.
  Interventions: Behavioral: Oral Hygiene instruction; Procedure: Dental Cleaning
- Control (No Intervention): Participants randomized to this arm will be instructed to continue with their usual oral hygiene practices for the duration of the study period.

INTERVENTIONS:
Behavioral: Oral Hygiene instruction — Participants will be instructed on the Modified Bass technique for toothbrushing: brushing with a soft bristled toothbrush held at a 45 degree angle to the gums and brushed in a circular motion. Participants will also be instructed to floss at least once per day using floss or another inter-dental device (e.g., floss pick).
  Arms: Participants receiving a dental cleaning and oral hygiene instruction
Procedure: Dental Cleaning — Participants will receive a dental cleaning according to the current standard of care for routine dental cleanings.
  Arms: Participants receiving a dental cleaning and oral hygiene instruction

SUMMARY:
This clinical trial is studying if bacteria found in a participant's bloodstream after brushing their teeth can be prevented with a dental cleaning and more education on how to best brush and care for their teeth. One group of participants will have a dental cleaning and oral health instructions and the other group of participants will not. Researchers will compare the blood test results from the two groups to see if the education made a difference in preventing bacteria and how long it stays in the bloodstream.

DETAILED DESCRIPTION:
This multi-center randomized clinical trial will determine if an intervention to improve oral hygiene and reduce gingival inflammation decreases the incidence and duration of bacteremia of Infective Endocarditis (IE) causing bacterial species, which may refocus longstanding guidelines on prevention for all people at risk for Infective Endocarditis (IE). The Standardized Brushing Hygienist will brush the participant's teeth over a 2-minute period, during and after which there will be 4 additional blood samples. The participant will then be randomized to an intervention or routine care group. The intervention will consist of a single session of tooth scaling and polishing, and oral hygiene instruction provided at the end of the Randomization Visit. Both groups will return for 3-week and 15-week visits, during which they will undergo a non-invasive oral examination and the brushing procedure with 5 blood samples (baseline and 4 additional blood samples after brushing begins). All blood samples will be cultured for bacteria of IE causing species.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Greater than 6 months since last dental hygiene prophylaxis (cleaning).
* 10 or more accessible teeth (including implants, with a minimum of 8 natural teeth).
* Willing and able to provide informed consent.
* Willing to comply with all study procedures and be available for the duration of the study.
* Willing to forgo routine professional dental cleanings while enrolled in the trial.

Exclusion Criteria:

* At high risk for IE, as defined by the 2007/2021 AHA Guidelines:
* Prosthetic cardiac valve or prosthetic material used for cardiac valve repair.
* Previous episode of IE.
* Cardiac transplantation recipient with cardiac valvulopathy.
* Specific congenital heart disease conditions.
* Pregnant, by self-report, or planning to become pregnant during the study period.
* Affected by a condition that, in the opinion of the investigator, may preclude them from study completion or put them at increased risk such as :
* Hemodialysis dependent.
* Have a long-term intravascular catheter (e.g., for chemotherapy or parenteral nutrition).
* Active injection drug use (IDU).
* Clotting disorder such as, hemophilia.
* Have a solid organ transplant or hematopoietic stem cell transplant, or ongoing treatment for hematologic cancer.
* Currently incarcerated.
* Systemic antibiotic use within the past 2 weeks.
* Undergoing orthodontic treatment with fixed appliances (brackets and wires) or plans to do so during the study period.
* Taking or requiring antibiotic prophylaxis prior to dental procedures for other reasons, e.g., to prevent prosthetic joint infection .
* Three or more teeth with moderate to severe gingival hyperplasia.
* Has clinically detectable emergent or urgent dental needs that, in the trained and calibrated Oral Examiner's opinion, would require definitive dental care during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2023-08-31 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of bacteremia | Baseline
  Blood samples are assessed for positivity of Infective Endocarditis (IE) causing oral species. A participant is defined as having bacteremia at a visit if that participant has at least one blood draw positive for bacteremia of IE-causing species during or after tooth brushing, provided that those IE-causing species were not present at the pre-brushing blood draw.
Incidence of bacteremia | Week 15
  Blood samples are assessed for positivity of Infective Endocarditis (IE) causing oral species. A participant is defined as having bacteremia at a visit if that participant has at least one blood draw positive for bacteremia of IE-causing species during or after tooth brushing, provided that those IE-causing species were not present at the pre-brushing blood draw.

SECONDARY OUTCOMES:
Change in Incidence of bacteremia | Baseline to Week 3
  Blood samples are assessed for positivity of Infective Endocarditis (IE) causing oral species. A participant is defined as having bacteremia at a visit if that participant has at least one blood draw positive for bacteremia of IE-causing species during or after tooth brushing, provided that those IE-causing species were not present at the pre-brushing blood draw.
Change in duration of bacteremia score | Baseline, Week 3, and Week 15
  At each visit, participants will have 5 blood samples drawn over the course of ~15 minutes. When a bacteremia occurs at a visit, its duration is defined as the last blood draw that tests positive for an IE-causing bacterial species that was not present at the pre-brushing draw. Possible values for duration are: 0 (no positive blood samples), 1 (only the blood draw during tooth brushing was positive), 2, 3, or 4, where the latter refer respectively to the subsequent blood samples.
Change in calculus index scores | Baseline, Week 3, and Week 15
  The calculus index, defined as the average calculus score (0 to 3 scale) from 4 sites per tooth on all teeth in the dentition, will be measured at each visit - Calculus will be assessed using the index of Ramfjord - 0 = absence of signs of inflammation; 1 = mild to moderate inflammatory gingival changes, not extending around the tooth; 2 = mild to moderately severe gingivitis extending all around the tooth; 3 = severe gingivitis characterized by- marked redness, swelling, tendency to bleed and ulceration - higher scores denote worse changes
Change in visible plaque scores | Baseline, Week 3, and Week 15
  The visible plaque score, defined as the percentage of surfaces with visible plaque across all teeth in the dentition, will be measured at each visit - Marginal dental plaque will be scored as visible or not visible using the criteria of Silness and Lӧe (1964) - Visible plaque corresponds to Silness and Lӧe scores of 2 and 3 - higher scores denote worse plaque
Change in gingival index scores | Baseline, Week 3, and Week 15
  The gingival index, defined as the average gingival score (0 to 3 scale) from 4 sites per tooth on all teeth in the dentition, will be measured at each visit - Gingivitis will be assessed using the Gingival Index of Lӧe and Silness - A score from 0.1-1.0 = mild inflammation; 1.1-2.0 = moderate inflammation from, and 2.1-3.0 signifies severe inflammation - higher scores denote increased inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lockhart, DDS, Principal Investigator — Wake Forest University Health Sciences
Locations (6):
- United States (6):
  - Tufts University School of Dental Medicine and Tufts University Health Sciences Campus, Boston, Massachusetts
  - University of Michigan School of Dentistry and Michigan Medicine, Ann Arbor, Michigan
  - Rutgers School of Dental Medicine, Newark, New Jersey
  - New York University, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Atrium Health's Carolinas Medical Center, Charlotte, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
A public use dataset will be available upon study completion.